CLINICAL TRIAL: NCT07252440
Title: A Prospective, International, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Evaluate the Efficacy and Safety of TTYP01 Tablets in Early Symptomatic Alzheimer's Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of TTYP01 Tablets in Early Symptomatic Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Auzone Biological Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTYP01-Ⅱ-AD
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: AD; Early Alzheimer's Disease
Keywords: AD; Alzheimer's Disease; TTYP01; Placebo-Controlled; Double-Blind; Early Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Experimental): 60 mg (2 TTYP01 30 mg tablets + 1 placebo tablet) BID
  Interventions: Drug: TTYP01 tables 60mg
- High-dose group (Active Comparator): 90 mg (3 TTYP01 30 mg tablets) BID
  Interventions: Drug: TTYP01 tables 90mg
- Placebo group (Placebo Comparator): 3 placebo tablets, BID
  Interventions: Drug: TTYP01 tables 0mg

INTERVENTIONS:
Drug: TTYP01 tables 60mg — 2 TTYP01 30 mg tablets + 1 placebo tablet BID
  Arms: Low-dose group
Drug: TTYP01 tables 90mg — (3 TTYP01 30 mg tablets
  Arms: High-dose group
Drug: TTYP01 tables 0mg — 3 placebo tablets
  Arms: Placebo group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled parallel Phase II core period study to evaluate the efficacy and safety of TTYP01 Tablets in early symptomatic AD (Mild cognitive impairment [MCI] due to AD, or mild AD dementia).

A total of 180 participants will be randomized into 3 parallel groups: 2 TTYP01 dose groups and 1 placebo group.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all the following criteria to be eligible for this study:

1. Age between 60 and 85 years (inclusive, based on the date of signing the informed consent), applicable to all genders.
2. Must meet the 2024 Alzheimer's Association (AA) Workgroup revised criteria for diagnosing MCI due to AD or mild AD dementia.
3. CDR score: At screening and baseline, the CDR global score must be 0.5 or 1.0, and the CDR memory score must be 0.5 or higher.
4. MMSE score: At screening, the MMSE score must be 22 or higher.
5. Body mass index (BMI): At screening, BMI must be greater than 17 and less than 35 (inclusive).
6. History of memory decline: A history of at least 6 months of gradual and progressive memory decline prior to signing ICF must be reported and confirmed by an informant.
7. Blood p-tau 217: positive (For participants with evidence suggesting Aβ-PET positivity, absence blood p-tau 217 determination is not considered a protocol deviation.).
8. Aβ- PET scan: Visual read of Aβ-PET scan must be positive.
9. Study partner: Must have a designated study partner who can support the participants and spend at least 8 h per week with them during the study. The partner must provide a separate written informed consent and be willing and able to provide follow-up information about the participant. They should regularly spend enough time with the participants to reliably meet study requirements. The study partner does not need to live with the participant but should be easily reachable during the study. If the partner is unable to continue supporting due to health or other reasons, it is allowed to replace with another eligible partner. The replacement partner must provide a separate written informed consent and be willing and able to provide follow-up information about the participant.
10. Concomitant medication: Participants who are receiving cholinesterase inhibitors and/or memantine for AD can be enrolled into the study, but must be on a stable dose for at least 12 weeks prior to baseline. For all other (i.e., non-AD-related) allowed concomitant medications, participants must receive a stable dose (not for topical, as needed [PRN], or discontinued medications) for at least 4 weeks prior to baseline unless otherwise stated.
11. Contraception:

    a.Male participants i.Male participants, regardless of childbearing potential, if their non-pregnant female partner is a female of childbearing potential, must agree to maintain abstinence (if this is their preferred and usual lifestyle) or to use a barrier method and another highly effective (failure rate less than 1%) method of contraception (see Section 17.5 for details) until 90 days after the last dose of IP.

    ii.Male participants with pregnant partners should use condoms during intercourse for the duration of the study and until the end of the estimated relevant potential exposure for women of childbearing potential (WOCBP; expected to be 90 days after the last dose of IP).

    iii.Male participants should refrain from sperm donation for the duration of the study and until 90 days following the last dose of IP.

    b.Female participants i.WOCBP must use, or be willing to use, two forms of effective contraception (a barrier method and one other highly effective method of contraception, as detailed in Section 17.5) during participation in the trial and for 90 days after the last dose of the IP.

    ii.WOCBP potential is defined as those who are:

    ① Following menarche

    ② From the time of menarche until becoming postmenopausal unless permanently sterile (see below) A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
    * In the absence of 12 months of amenorrhea, confirmation with more than one follicle-stimulating hormone (FSH) measurement is required.
    * Individuals receiving hormone replacement therapy (HRT) whose menopausal status is in doubt will be required to use a non-estrogenic, highly effective contraceptive method if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment.

    Permanent sterilization methods and gender-affirming procedures (for the purpose of this study) include:
    * Documented hysterectomy
    * Documented bilateral salpingectomy
    * Documented bilateral oophorectomy
    * For individuals with permanent infertility due to an alternate medical cause other than the above, (e.g., Mullerian agenesis, androgen insensitivity, gonadal dysgenesis), investigator discretion should be applied to determining study entry.

    iii.All WOCBP must be negative at Visit 1 based on a serum pregnancy test.
12. Informed consent: Must obtain a voluntary signed ICF, approved by an Ethics Committee, from the participants or their legal representative before any study procedure.
13. Language proficiency: Must be fluent in the language used at the study site.
14. Protocol compliance: Must be willing and able to comply with all aspects of the protocol.

Exclusion Criteria

Participants who meet any of the following exclusion criteria will not be eligible for the study:

1. History of intracranial infection or traumatic brain injury.
2. Severe coronary heart disease, cardiac insufficiency (New York Heart Association Class Ⅲ and Class IV), atrial fibrillation, and other heart diseases within six months prior to signing ICF.
3. Malignancy:

   * History of cancer within the last 3 years, with the exception of non-metastatic basal and/or squamous cell carcinoma of the skin, in situ cervical cancer, nonprogressive prostate cancer, or other cancers with a low risk of recurrence or spread.
   * Intracranial space occupying lesions or brain tumors will be excluded unless, based on the opinion of the investigators and medical monitors, the medical condition will not interfere with cognitive assessments and safety.
4. Severe hematologic disorders, such as myelodysplastic syndrome, aplastic anemia, lymphoma, leukemia, etc.
5. Peptic ulcer or obstruction or other diseases that affect the absorption of oral medication.
6. Any neurological disorder that may cause cognitive impairment beyond the impact of AD.
7. Any psychiatric diagnosis or neuropsychiatric symptom (such as hallucinations, major depression, or delusions) that may interfere with the participant's study procedure.
8. A history of transient ischemic attack (TIA), stroke, or seizure in the 12 months prior to signing ICF.
9. The Hachinski Ischemic Index Scale (HIS) at screening > 4 points.
10. ECG at screening or at baseline showing prolonged QTcF [Fridericia correction formula, see Section 17.4] (QTcF > 480 ms in women; QTcF > 470 ms in men) or other clinically significant abnormalities of the ECG that are considered by the investigator to be unsuitable for participation in a clinical study (e.g., heart rate < 50 beats/min, sinus node lesions, Morse II or third-degree atrioventricular block, etc.).
11. The Geriatric Depression Scale (GDS) score at screening ≥ 8 points.
12. Contraindications to MRI scans, including pacemakers/defibrillators, ferromagnetic metal implants (in addition to those approved for safe use in MRI scanners, such as cranial and cardiac devices).
13. Contraindications with PET scanning, allergies to tracers.
14. Brain MRI at screening reveals evidence of other clinically significant lesions, suggesting a possible diagnosis of dementia other than AD.
15. Brain MRI at screening reveals the presence of a single hemorrhage with a maximum diameter > 10 mm and investigator assesses the participant is unsuitable for this study; Evidence of angioedema.
16. Participants with inadequately controlled bleeding disorder (including platelet count < 100,000/µL or international normalized ratio [INR] > 1.5).
17. Thyroid stimulating hormone levels above or below the normal range. Participants with results of other thyroid function tests that fall outside the normal range will be excluded only if they are considered clinically significant by the investigator.
18. Laboratory test results for serum vitamin B12 levels below the normal range, as well as participants who are receiving vitamin B12 supplement therapy.
19. Positive serological finding for human immunodeficiency virus (HIV), active syphilis, Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV) antibody.
20. Any other clinically significant abnormalities in physical examination, vital signs, laboratory tests, or ECG present at screening or baseline that the investigator determines the situations that affected the safety of the participants or other interferences with the study.
21. Have a known or suspected history of drug or alcohol abuse.
22. Serious or unstable disease, or any other medical condition (e.g., heart, respiratory, gastrointestinal, liver, kidney, endocrine and nervous system disease, including poorly controlled hypertension, with a systolic blood pressure of ≥160mmHg or a diastolic blood pressure of ≥100 mmHg; Poorly controlled diabetes, etc.) that the investigator believes may affect the participant's safety or interfere with study evaluation.
23. Previous use of prohibited drugs, including disease-modifying drugs (Such as approved lecanemab, donemab, etc. or other disease-modifying investigational medicinal products), anti-oxidative stress drugs (other formulations of edaravone).
24. Have scheduled surgical procedures requiring general anesthesia during the study period. For a scheduled procedure that requires only local anesthesia and performed as a day procedure without the need for post-operative hospitalization, participant does not need to be excluded if the investigator determines that the procedure does not interfere with study procedures or participant safety.
25. Severe vision, hearing, reading, comprehension, or physical dysfunction that prevents the participant from accurately performing neuropsychological tests.
26. Have been diagnosed with serious active liver disease, such as acute hepatitis, chronic active hepatitis, cirrhosis, etc., or alanine transaminase (ALT) > 2 × upper limit of normal (ULN) or aspartate aminotransferase (AST) > 2 × ULN, or total bilirubin (TBIL) > 1.5 × ULN.
27. Have been diagnosed with severe active kidney disease, renal insufficiency; or serum creatinine > 1.5 × ULN or creatinine clearance < 50 mL/min at screening and baseline (Calculated based on the Cockcroft-Gault formula, see Section 17.6 for details).
28. Have severe systemic disease and life expectancy is < 2 years.
29. Answer "yes" to C-SSRS suicidal ideation Type 4 or 5, or any suicidal behavior assessment within 6 months before screening, at screening, or at the baseline visit, or has been hospitalized or treated for suicidal behavior in the past 5 years before screening.
30. Allergic to edaravone, sodium bisulfite, or soluplus excipients (Note: Asthma patients are sensitive to sulfites and may have allergic reactions. For patients with a history of asthma, the investigator will carefully assess whether to enroll them.).
31. History of major surgery within 4 weeks prior to enrollment.
32. Have participated in, or are currently participating in, another clinical study within the 30 days prior to randomization (Participants who have previously participated in clinical studies of disease-modifying drugs targeting Aβ and/or tau pathology will follow exclusion criteria 23).
33. Participants who have received cholinesterase inhibitors, memantine within 12 weeks prior to randomization and stopped treatment due to safety concerns or other reasons and refuse to or unable to receive it again.
34. Female participants who are pregnant, breastfeeding, planning to become pregnant recently, or unwilling to use contraceptive measures.
35. Have other conditions that investigator believes the participant is unsuitable for this study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2028-10-23 (Estimated); Study Completion 2028-11-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) score at Week 78. | Baseline to Week 78
Number of participants with Adverse events, serious adverse events, adverse events of special interest | Baseline to Week 78

SECONDARY OUTCOMES:
TTYP01 PK parameter (AUC (0-t,0-24,∞) | 78 weeks
Change From Baseline in Amyloid Positron Emission Tomography (PET) Using Centiloids at Week 39 and Week 78 | Baseline to Week 39 and Week78
Change from baseline in blood p-tau 217 at week 78. | baseline to week 78
Changes from baseline in Mini-Mental State Examination (MMSE). | Week 13, 26, 39, 52, 65, and 78
Change from Baseline in Alzheimer Disease Assessment Scale - Cognitive Subscale 13 (ADAS-cog13) at Week 39 and Week 78. | baseline to week 39 and week 78

OTHER OUTCOMES:
To explore the exposure-clinical effect relationship of TTYP01 Tablets in treating early symptomatic AD. | week78
  Correlation analyses between edaravone exposure in blood and changes of CDR-SB, ADCOMS, ADAS-Cog13, ADCS-ADL, and MMSE score at Week 78.
To explore the exposure-effect relationship of TTYP01 Tablets on cerebral amyloid plaque deposition, and MRI brain volume. | week39 ,week78
  Correlation analyses between edaravone exposure in blood and changes of Aβ-PET and MRI brain volume at Week 39 and Week 78.
To assess the effect of TTYP01 vs. placebo on clinical progression, behavioral, neuropsychiatric symptom and study partner burden in early symptomatic AD patients. | Week 13, 26, 39, 52, 65, and 78.
  The proportion of clinical progression or clinical improvement in the test group compared with the placebo group at Week 13, 26, 39, 52, 65, and 78.
  ①Progression criteria: 1. Any increase in the overall Clinical Dementia Rating Scale (CDR) score from baseline; 2. CDR-SB is higher than baseline. Criteria 1 and 2 are evaluated separately.
  ②Improvement criteria: 1. Any decrease in the overall CDR score from baseline; 2. CDR-SB is lower than baseline. Criteria 1 and 2 are evaluated separately.
  Time to clinical progression (criteria 1: time to increase in overall CDR score from baseline; 2: time to increase in CDR-SB from baseline).
  Changes in Neuropsychiatric Inventory (NPI) scores from baseline at Week 26, 52 and 78.
  Changes from baseline in the Zarit Burden Interview (ZBI) at Week 26, 52, and 78.
To evaluate the effects of TTYP01 Tablets on blood PD markers (AD biomarkers and cytokines). | Week 4, 8, 13, 39 and 78.
  Changes from baseline in levels of AD biomarkers amyloid-beta peptides (Aβ42/40), Glial Fibrillary Acidic Protein (GFAP), and neurofilament light chain (NfL) at Week 4, 8, 13, 39 and 78.
  Changes in cytokines: interferon-gamma (IFN-γ), interleukin-1β (IL-1β), interleukin-6 (IL-6) and tumor necrosis factor-α (TNF-α) at Week 4, 8, 13, 39 and 78
To evaluate the relationship between brain amyloid levels and blood biomarkers (including but not limited to blood p-tau 217, Aβ42/40, NfL, GFAP, and cytokines (IFN-γ, IL-1β, IL-6 and TNF-α) in participants with AD. | week39,week78
  Correlation between changes in brain amyloid levels (Aβ-PET), and changes in blood biomarkers (including but not limited to blood p-tau 217, Aβ42/40, NfL, GFAP and cytokines (IFN-γ, IL-1β, IL-6 and TNF-α).
To evaluate the relationship between volume MRI (vMRI) and clinical changes (CDR-SB, ADCOMS, ADAS-Cog13, ADCS-ADL and MMSE) in participants with AD. | week78
  Correlation between clinical changes (CDR-SB, ADCOMS, ADAS-Cog13, ADCS-ADL, and MMSE) and changes in vMRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital., Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No